CLINICAL TRIAL: NCT05012397
Title: A Phase 2 Basket Study of Milademetan in Advanced/Metastatic Solid Tumors (MANTRA-2)
Brief Title: Milademetan in Advanced/Metastatic Solid Tumors
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Rain Oncology Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RAIN-3202
Record Dates: First submitted 2021-08-13; First posted 2021-08-19 (Actual); Results first posted 2024-10-17 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Solid Tumors; Head and Neck Carcinoma; Cholangiocarcinoma; Sarcoma; Lung Adenocarcinoma; Bladder Urothelial Carcinoma; Stomach Adenocarcinoma; Breast Cancer Invasive; Ovarian Carcinoma; Cervical Cancer; Non Small Cell Lung Cancer; Gastric Cancer; Biliary Tract Cancer; Melanoma; Pancreas Cancer; MDM2 Gene Amplification; Testicular Germ Cell Tumor; Adrenocortical Carcinoma
Keywords: MDM2; Milademetan; Basket Study
MeSH Terms: conditions — Cholangiocarcinoma; Sarcoma; Adenocarcinoma of Lung; Ovarian Neoplasms; Uterine Cervical Neoplasms; Carcinoma, Non-Small-Cell Lung; Stomach Neoplasms; Biliary Tract Neoplasms; Melanoma; Pancreatic Neoplasms; Testicular Germ Cell Tumor; Adrenocortical Carcinoma | interventions — milademetan

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Milademetan (RAIN-32) (Experimental): 260 mg once dailly orally on Days 1 to 3 and Days 15 to 17 of each 28-day cycle
  Interventions: Drug: RAIN-32

INTERVENTIONS:
Drug: RAIN-32 — 260 mg once daily orally on Days 1 to 3 and Days 15 to 17 of each 28-day cycle
  Other Names: Milademetan

SUMMARY:
Phase 2, multicenter, single-arm, open-label basket study designed to evaluate the safety and efficacy of milademetan in patients with advanced or metastatic solid tumors refractory or intolerant to standard-of-care therapy that exhibit wild-type (WT) TP53 and MDM2 copy number (CN) ≥ 8 using prespecified biomarker criteria.

DETAILED DESCRIPTION:
Approximately 65 patients will be enrolled to receive milademetan.

Patients will receive the study drug until reaching unequivocal disease progression (per Response Evaluation Criteria in Solid Tumors [RECIST] version [v]1.1), as determined by the Investigator; experiencing unmanageable toxicity; or until other treatment discontinuation criteria are met. Patients may be treated beyond tumor progression if they are experiencing clinical benefit based on the assessment of the Investigator in discussion with the Medical Monitor.

All patients will be followed for documentation of disease progression and survival information (i.e., date and cause of death). Long-term follow-up will continue every 12 weeks (± 7 days) until the endpoint of death, the patient is lost to follow-up, or for 24 months following the final dose of the study drug, whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

* Histologically and/or cytologically confirmed diagnosis of a cancer that is a locally advanced or metastatic solid tumor
* Measurable tumor lesion(s) in accordance with RECIST v1.1
* Received all standard therapy appropriate for their tumor type and stage of disease or, in the opinion of the Investigator, would be unlikely to tolerate or derive clinically meaningful benefit from appropriate standard-of-care therapy
* Resolution of any clinically relevant toxic effects of prior chemotherapy, surgery, radiotherapy, or hormonal therapy
* Presence of WT TP53 and MDM2 gene amplification by tumor tissue/blood testing, defined as ≥ 8 copies in tumor tissue by central laboratory or ≥ 8 copies or 4-fold increase in tumor tissue or blood by local testing
* Prescreening for TP53 and MDM2 at a Central Laboratory:

  * MDM2 amplification: CN unknown and where CN cannot be derived for documentation by interpretation of reported results
  * MDM2 amplification: CN 6 to 7.9
  * MDM2 amplification: 3-3.9-fold increase
  * MDM2 amplification with CN ≥ 8 and with equivocal TP53 mutation upon discussion with Sponsor's Medical Monitor
* ECOG performance status of 0 or 1
* Adequate bone marrow function:

  * Platelet count ≥ 100 × 10^9/L
  * Hemoglobin ≥ 9.0 g/dL
  * Absolute neutrophil count ≥ 1.5 × 10^9/L
* Adequate renal function

  * Creatinine clearance ≥ 30mL/min, as calculated using the modified Cockcroft-Gault equation
* Adequate hepatic function

  * Alanine aminotransferase and aspartate aminotransferase ≤ 3 × upper limit of normal (ULN) if no liver metastases are present; ≤ 5 × ULN if liver metastases are present
  * Total bilirubin ≤ 1.5 × ULN, or ≤ 3 x ULN in the presence of liver metastases

Exclusion Criteria:

* Prior treatment with a murine double minute 2 (MDM2) inhibitor
* Well-differentiated/dedifferentiated liposarcoma or intimal sarcoma/cardiac sarcoma
* Primary malignancies that required systemic antineoplastic treatment within the previous 2 years, except for localized cancers that have apparently been cured
* Has a primary malignant brain tumor of any grade or histology
* Untreated brain metastases
* Gastrointestinal conditions that could affect the absorption of milademetan, in the opinion of the Investigator
* Known HIV infection or active hepatitis B or C infection
* Major surgery ≤ 3 weeks of the first dose of milademetan
* Curative-intent radiation therapy ≤ 4 weeks or palliative radiation therapy
* Uncontrolled or significant cardiovascular disease

  1. QTcF at rest, where the mean QTcF interval is > 480 milliseconds
  2. Myocardial infarction within 6 months
  3. Uncontrolled angina pectoris within 6 months
  4. New York Heart Association Class 3 or 4 congestive heart failure
  5. Uncontrolled hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-10-15 (Actual); Study Completion 2023-10-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - Stanford University Medical Center, Palo Alto, California
  - Florida Cancer Specialists, Fort Myers, Florida
  - Florida Cancer Specialists, St. Petersburg, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Hematology Oncology Associates of Central NY, Syracuse, New York
  - Duke University Medical Center, Durham, North Carolina
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Sanford Health, Sioux Falls, South Dakota
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - Northwest Medical Specialities, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gounder MM, Bauer TM, Schwartz GK, Weise AM, LoRusso P, Kumar P, Tao B, Hong Y, Patel P, Lu Y, Lesegretain A, Tirunagaru VG, Xu F, Doebele RC, Hong DS. A First-in-Human Phase I Study of Milademetan, an MDM2 Inhibitor, in Patients With Advanced Liposarcoma, Solid Tumors, or Lymphomas. J Clin Oncol. 2023 Mar 20;41(9):1714-1724. doi: 10.1200/JCO.22.01285. Epub 2023 Jan 20. PMID 36669146

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All enrolled participants (40 participants) received the study medication. Twenty-eight (28) discontinued treatment. Fourteen (14) completed the study.
Groups:
- Milademetan (RAIN-32): 260 mg once daily (QD) orally on Days 1 to 3 and Days 15 to 17 of each 28-day cycle
Period: Overall Study
Arm/Group | Milademetan (RAIN-32)
Started | 40
Completed | 14
Not Completed | 26
Not completed — Death | 10
Not completed — Physician Decision | 9
Not completed — Withdrawal by Subject | 5
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Arm/Group | Milademetan (RAIN-32)
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.5 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 32
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Number; unit: participants]
  United States | 40
BMI [Mean (Standard Deviation); unit: kg/m2] | 24.8 (5.1)

OUTCOME MEASURES:

1. Primary Outcome: To Determine the ORR of Treatment With Milademetan in Patients With Advanced/Metastatic Solid Tumors With MDM2 Gene Amplification.
Description: Overall Response Rate (ORR) of treatment with milademetan, as defined as the percentage of patients who have achieved confirmed complete response (CR) or Partial Response (PR) according to RECIST v1.1
Time Frame: From first dose date to first confirmed complete or partial response or study completion date; up to 23.5 months.
Population: This analysis is conducted in all participants within the Centrally confirmed population (CCP) which is defined as all participants who had at least one dose of study treatment and also have WT TP53 and MDM2 amplification with CN ≥ 8 by central testing.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Milademetan (RAIN-32)
Number analyzed (Participants) | 31
percentage of participants | 3.2 [0.1 to 16.7]

2. Secondary Outcome: Duration of Response (DOR)
Description: DOR defined as the time from the date of first documentation of CR or PR according to RECIST v1.1 to the date of disease progression or death due to any cause according to Investigator assessment
Time Frame: From start date of response to first PD or study completion date; up to 23.5 months
Population: This analysis is conducted in all participants within the Centrally confirmed population (CCP) who had a confirmed CR or PR.
Measure: Number; unit: months
Arm/Group | Milademetan (RAIN-32)
Number analyzed (Participants) | 1
months | 3.84

3. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS defined as the time from the date of the first dose of the study drug to the earliest date of the first objective documentation of radiographic disease progression or death due to any cause according to Investigator assessment
Time Frame: From the first dose date to the earliest date of recurrence, progression, death, or study completion; up to 23.5 months
Population: The efficacy analysis is conducted in all participants within the Centrally confirmed population (CCP).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Milademetan (RAIN-32)
Number analyzed (Participants) | 31
months | 3.5 [1.8 to 3.7]

4. Secondary Outcome: Growth Modulation Index (GMI)
Description: GMI defined as the ratio of Time to Progression (TTP) with the nth line of therapy (TTPn; here defined as milademetan) to the most recent prior line of therapy (TTPn-1)
Time Frame: From the start date of the most recent prior line of therapy to the PD date on the study; up to 23.5 months
Population: The efficacy analysis is conducted in all participants within the Centrally confirmed population (CCP).
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Milademetan (RAIN-32)
Number analyzed (Participants) | 31
months | 0.76 [0.47 to 0.98]

5. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR defined as the percentage of patients with confirmed CR, PR, or stable disease (SD) for ≥ 16 weeks
Time Frame: From first dose date to first CR, PR, or stable disease (SD) >= 16 weeks, or study completion date; up to 23.5 months
Population: The efficacy analysis is conducted in all participants within the Centrally confirmed population (CCP).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Milademetan (RAIN-32)
Number analyzed (Participants) | 31
percentage of participants | 22.6 [9.6 to 41.1]

ADVERSE EVENTS:
Time Frame: From the first dose date to 30 days after the last dose date or study completion date whichever came first; up to 23.5 months
Description: meets definition
Arm/Group | Milademetan (RAIN-32)
All-Cause Mortality (participants affected / at risk) | 10/40
Serious Adverse Events (participants affected / at risk) | 11/40
Other Adverse Events (participants affected / at risk) | 40/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Milademetan (RAIN-32) (N=40)
Anemia (Blood and lymphatic system disorders) | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 3
Leukocytosis (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Normocytic anemia (Blood and lymphatic system disorders) | 1
Dizziness (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Gastric haemorrhage (Gastrointestinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Tympanic membrane perforation (Ear and labyrinth disorders) | 1
blood creatine increased (Investigations) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Tumor Haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Milademetan (RAIN-32) (N=40)
Thrombocytopenia (Blood and lymphatic system disorders) | 21
vomiting (Gastrointestinal disorders) | 20
Nausea (Gastrointestinal disorders) | 18
Fatigue (General disorders) | 16
Diarrhoea (Gastrointestinal disorders) | 13
Anemia (Blood and lymphatic system disorders) | 10
Neutropenia (Blood and lymphatic system disorders) | 9
Abdominal pain (Gastrointestinal disorders) | 8
Ascites (Gastrointestinal disorders) | 5
Dizziness (Nervous system disorders) | 5
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5
Back pain (Musculoskeletal and connective tissue disorders) | 4
Decreased appetite (Metabolism and nutrition disorders) | 4
Headache (Nervous system disorders) | 4
Hypophosphatemia (Metabolism and nutrition disorders) | 4
Edema peripheral (General disorders) | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4
Pruritus (Skin and subcutaneous tissue disorders) | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
COVID-19 (Respiratory, thoracic and mediastinal disorders) | 3
Constipation (Gastrointestinal disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Dry mouth (Gastrointestinal disorders) | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 3
Hypokalaemia (Metabolism and nutrition disorders) | 3
Influenza (Infections and infestations) | 3
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3
Pyrexia (General disorders) | 3
Blood Creatinine increased (Investigations) | 2
Dysgeusia (Nervous system disorders) | 2
Face oedema (General disorders) | 2
Hyponatraemia (Metabolism and nutrition disorders) | 2
Mucosal inflammation (General disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Seizure (Nervous system disorders) | 2
Taste disorder (Nervous system disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-11-21): https://cdn.clinicaltrials.gov/large-docs/97/NCT05012397/Prot_000.pdf
  • Statistical Analysis Plan (2023-10-28): https://cdn.clinicaltrials.gov/large-docs/97/NCT05012397/SAP_001.pdf